CLINICAL TRIAL: NCT02941016
Title: Vascular Inflammation and Cholesterol Lowering Therapy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Logistic reasons
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Rasmus S. Ripa, Staff Physician, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0002
Record Dates: First submitted 2016-10-18; First posted 2016-10-21 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Lipid Lowering, Vascular Inflammation
MeSH Terms: interventions — evolocumab; alirocumab

ARMS (1):
- Lipid lowering (Experimental)
  Interventions: Drug: Evolocumab or Alirocumab

INTERVENTIONS:
Drug: Evolocumab or Alirocumab — All patients are treated with PCSK-9 inhibitors (Evolocumab or Alirocumab) to lower cholesterol

SUMMARY:
This study aim to detect change in vascular inflammation following intense lipid lowering therapy

ELIGIBILITY:
Inclusion Criteria:

* treatment with PCSK-9 inhibitors

Exclusion Criteria:

* Infection Pregnancy Severe claustrophobia Weight >140 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2020-10 (Estimated); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Change in vascular inflammation | 12 weeks
  Change in standard uptake value (SUV) of flourdeoxyglucose (FDG) before and after initiation of lipid lowering therapy

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus S Ripa, MD, DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark